CLINICAL TRIAL: NCT01212406
Title: A Randomized Double Blind Placebo Controlled Trial With Vitamin D to Prevent Bronchiolitis Obliterans Syndrome After Lung Transplantation
Brief Title: Vitamin D in Bronchiolitis Obliterans Syndrome
Acronym: VIT001
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIT001
Record Dates: First submitted 2010-09-28; First posted 2010-09-30 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2013-10

CONDITIONS: Allograft Rejection; Lung Transplantation; Bronchiolitis Obliterans
Keywords: Organ rejection; Lung transplantation; Bronchiolitis Obliterans; Vitamin D; Prevention
MeSH Terms: conditions — Bronchiolitis Obliterans | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Olive oil
  Interventions: Drug: Vitamin D
- Vitamin D (Experimental): Addition of D-cure (100.000U) to standard care
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Every month 100.000 units of vitamin D in syringe Exacta-Med Oral Dispenser during 2 years and re-evaluation after 3 years
  Other Names: D-Cure

SUMMARY:
Vitamin D deficiency occurs in around 50% of our transplant population. Preventive treatment with Vitamin D (D-cure) can reduce the prevalence of Bronchiolitis Obliterans Syndrome after lung transplantation

DETAILED DESCRIPTION:
* Prospective, interventional, randomized, double-blind, placebo-controlled trial.
* Clinical setting (tertiary University Hospital).
* Investigator-driven, no pharmaceutical sponsor.
* Lung transplant recipients.
* Add-on of study-drug (placebo or vitamin D) to 'standard of care' (standardized, routine immunosuppressive and infectious prophylactic protocol).
* 1:1 inclusion ratio (placebo:Vitamin D).
* Randomisation at discharge after informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Stable LTx recipients at discharge after transplantation.
* Signed informed consent
* Adult (age at least 18 years old at moment of transplantation)
* Able to take oral medication

Exclusion Criteria:

* Prolonged and/or complicated Intensive care unit-course after transplantation.
* Early (<30 days post-transplant) post-operative death
* Major suture problems (airway stenosis or stent)
* Retransplantation (lung)
* Previous transplantation (solid organ)
* Multi-organ transplantation (lung+ other solid organ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of Bronchiolitis Obliterans syndrome (BOS) (grade 1) at 2 years after transplantation | 2 years after transplantation
  BOS= decline in forced expiratory volume in 1 second (FEV1) with at least 80% compared to the best post-operative value
Prevalence of BOS (grade 1) at 3 years after transplantation | 3 years after transplantation
  her-evaluation of data

SECONDARY OUTCOMES:
Bronchoalveolar lavage | during 2 and 3y of follow-up
  cellularity, protein and mRNA concentration and microbiology
Peripheral blood | During 2 and 3 years of follow-up
  Protein and mRNA concentration, cellularity
Rejection rates | During 2 and 3 years of follow-up
  Acute rejection and lymphocytic bronchiolitis rates
Reflux | During 2 and 3 years of follow-up
  clinical and biochemical approach
Infection rates | During 2 and 3 years of follow-up
  cytomegalovirus (CMV) and non- CMV infection rates

CONTACTS AND LOCATIONS:
Overall Officials: Geert M Verleden, MD, PhD, Principal Investigator — UZ gasthuisberg
Locations (1):
- UZ Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Ramirez AM, Wongtrakool C, Welch T, Steinmeyer A, Zugel U, Roman J. Vitamin D inhibition of pro-fibrotic effects of transforming growth factor beta1 in lung fibroblasts and epithelial cells. J Steroid Biochem Mol Biol. 2010 Feb 15;118(3):142-50. doi: 10.1016/j.jsbmb.2009.11.004. Epub 2009 Nov 17. PMID 19931390
- [Background] Zittermann A, Schleithoff SS, Gotting C, Fuchs U, Kuhn J, Kleesiek K, Tenderich G, Koerfer R. Calcitriol deficiency and 1-year mortality in cardiac transplant recipients. Transplantation. 2009 Jan 15;87(1):118-24. doi: 10.1097/TP.0b013e31818c2708. PMID 19136901
- [Background] Janssens W, Bouillon R, Claes B, Carremans C, Lehouck A, Buysschaert I, Coolen J, Mathieu C, Decramer M, Lambrechts D. Vitamin D deficiency is highly prevalent in COPD and correlates with variants in the vitamin D-binding gene. Thorax. 2010 Mar;65(3):215-20. doi: 10.1136/thx.2009.120659. Epub 2009 Dec 8. PMID 19996341
- [Background] Vanaudenaerde BM, Meyts I, Vos R, Geudens N, De Wever W, Verbeken EK, Van Raemdonck DE, Dupont LJ, Verleden GM. A dichotomy in bronchiolitis obliterans syndrome after lung transplantation revealed by azithromycin therapy. Eur Respir J. 2008 Oct;32(4):832-43. doi: 10.1183/09031936.00134307. PMID 18827151
- [Background] Estenne M, Maurer JR, Boehler A, Egan JJ, Frost A, Hertz M, Mallory GB, Snell GI, Yousem S. Bronchiolitis obliterans syndrome 2001: an update of the diagnostic criteria. J Heart Lung Transplant. 2002 Mar;21(3):297-310. doi: 10.1016/s1053-2498(02)00398-4. No abstract available. PMID 11897517